CLINICAL TRIAL: NCT00051974
Title: A Randomized, Multicenter, Open-Label, Phase 2 Study of VELCADE Alone or VELCADE Plus Docetaxel in Previously Treated Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Phase 2 Study of VELCADE Alone or VELCADE® Plus Docetaxel in Previously Treated Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M34102-048
Record Dates: First submitted 2003-01-21; First posted 2003-01-22 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-02

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bortezomib; WW Domain-Containing Oxidoreductase

INTERVENTIONS:
Drug: VELCADE™ (bortezomib) for Injection (formerly PS-341)

SUMMARY:
The purpose of this study is to evaluate how tumors in patients with non-small cell lung cancer respond to treatment with VELCADE alone versus VELCADE given with docetaxel and also to see what effects (good and bad) it has on you and your cancer.

DETAILED DESCRIPTION:
In this study, patients with non-small cell lung cancer that is no longer responding to standard medical treatment with another anti-cancer drug will be randomly chosen to receive treatment with VELCADE alone or VELCADE in combination with docetaxel. Patients have almost equal chance of getting into either of the two treatment arms listed above.

ELIGIBILITY:
Inclusion Criteria

* Inoperable, locally advanced (Stage IIIB) or metastatic (Stage IV) NSCLC that has been histologically or cytologically confirmed.
* No more than 1 prior chemotherapy regimen.
* 18 years of age or older.
* Measurable or evaluable disease.
* KPS ≥70%.
* Life expectancy greater than 3 months.
* Female patient is either post-menopausal, surgically sterilized, or willing to use an acceptable method of birth control for the duration of the study.
* Male patient agrees to use an acceptable method of birth control for the duration of the study.
* Provide written informed consent before any study-related procedure not part of normal medical care is conducted.
* Willing and able to comply with the protocol requirements.

Exclusion Criteria

* Peripheral neuropathy of Grade 2 or greater intensity, as defined by the NCI Common Toxicity Criteria (CTC):

  * Grade 2: Objective sensory loss or paresthesia (including tingling), interfering with function, but not interfering with activities of daily living (ADLs).
  * Grade 3: Sensory loss or paresthesia interfering with ADLs.
  * Grade 4: Permanent sensory loss that interferes with function.
* Previous treatment with VELCADE.
* Previous treatment with docetaxel (prior treatment with paclitaxel will be allowed).
* Chemotherapy within 4 weeks prior to enrollment.
* Radiation therapy within 4 weeks prior to enrollment.
* Monoclonal antibodies within 6 weeks prior to enrollment.
* Any major surgery within 4 weeks prior to enrollment.
* Inadequate organ function at the Screening visit as defined by the following laboratory values:

  * Platelet count ≤100,000 x 109/L
  * Hemoglobin ≤8.0 g/dL
  * Absolute neutrophil count (ANC) ≤1.5 x 109/L
  * Aspartate transaminase (AST) ≥3 x the upper limit of the normal range (ULN)
  * Alanine transaminase (ALT) ≥3 times ULN
  * Creatinine ≥1.8 mg/dL
  * Total bilirubin ≥2 times ULN
* Myocardial infarction within 6 months prior to enrollment or has New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* No history of brain metastases or central nervous system disease.
* Active systemic infection requiring treatment.
* Treatment for a cancer other than NSCLC within 5 years prior to enrollment, with the exception of basal cell carcinoma or cervical cancer in situ.
* History of allergic reaction attributable to compounds containing boron or mannitol.
* Known to be human immunodeficiency virus (HIV)-positive. Patients assessed by the investigator to be at risk for HIV infection should be tested in accordance with local regulations.
* Known to be hepatitis B surface antigen-positive or has known active hepatitis C infection. Patients assessed by the investigator to be at risk for hepatitis B or C infection should be tested in accordance with local regulations.
* Poorly controlled hypertension, diabetes mellitus, or another serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Pregnant or breast-feeding female patient. Confirmation that the patient is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during the Screening period. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Currently enrolled in another clinical research study or has received an investigational agent for any reason within 4 weeks of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155
Dates: Start 2002-12; Primary Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - U of Alambama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Cedars-Sinai Comprehensive Cancer Center, Los Angeles, California
  - UCLA Medical Center Thoracic Malignancy, Los Angeles, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Univeristy of Florida Shands Cancer Center, Gainesville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Atlanta VAMC, Decatur, Georgia
  - Mass. General Hospital Hem/Onc. Associates, Boston, Massachusetts
  - DBA Kansas City Cancer Centers, Kansas City, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Washington University, Barnard Cancer Center, St Louis, Missouri
  - Carolinas Hematology-Oncology Associates, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Kimmel Cancer Center at Jefferson, Philadelphia, Pennsylvania
  - Vanderbilt University-Clinical Trials Center, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Hunstman Cancer Institute-University of Utah, Salt Lake City, Utah
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin